CLINICAL TRIAL: NCT06480110
Title: Ebastine in Combination With Docetaxel as a Treatment for Castration-resistant Metastatic Prostate Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Danish Cancer Society (Other)
Responsible Party: Principal Investigator, Helle Pappot, Professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ebas0001
Record Dates: First submitted 2020-11-18; First posted 2024-06-28 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
MeSH Terms: interventions — Docetaxel; ebastine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Standard docetaxel (10 cycles) plus ebastine daily
  Interventions: Drug: Docetaxel + Ebastine
- Comparator (Active Comparator): Standard docetaxel (10 cycles) without ebastine
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Docetaxel + Ebastine — Ebastine is administered once daily.
  Other Names: Kestine (Ebastine)
  Arms: Intervention
Drug: Docetaxel — docetaxel every three weeks
  Arms: Comparator

SUMMARY:
This is an open-label phase I/II study evaluating the addition of ebastine to docetaxel in the treatment for metastatic castration resistant prostate cancer.

Patients will be randomized in a 2:1 fashion to receive ebastine daily during and after treatment with a maximum of 10 courses of docetaxel.

The primary endpoint is change in the profile of urinary and blood lipids to indicate absorption and possible efficacy of ebastine.

Secondary endpoints include PSA response and radiologic progression free survival.

DETAILED DESCRIPTION:
The complete study protocol can be studied by contacting the authors.

ELIGIBILITY:
Inclusion Criteria:

* 1. Have a histologically confirmed adenocarcinoma or poorly differentiated carcinoma of the prostate (carcinomas with pure small-cell histology or pure high grade neuroendocrine histology are excluded; neuroendocrine differentiation is allowed).

  2. Surgically or medically castrated, with serum testosterone levels of ≤ 50 ng/dL equivalent to 1.7 nmol/L. For patients, currently being treated with luteinizing hormone-releasing hormone (LHRH) agonists, i.e., patients who have not undergone an orchiectomy, therapy must be continued throughout the study.

  3. Have evidence of disease progression after prior therapy for mCRPC:

Disease progression after initiation of most recent therapy is based on any of the following criteria:

* Rise in PSA: a minimum of 2 consecutive rising levels, with an interval of ≥ 1 week between each determination. The most recent screening measurement must have been ≥ 2 ng/mL
* Transaxial imaging: new or progressive soft tissue masses on CT or MRI scans as defined by RECIST 1.1
* Radionuclide bone scan: at least 2 new metastatic lesions 4. Signed informed consent obtained prior to initiation of any study-specific procedures or treatment 5. Age ≥ 18 years 6. Life expectancy ≥ 3 months 7. Performance status 0 - 1 8. Adequate organ functions

  1. Hematological: absolute neutrophil count (ANC) >1.5 x 109/L, platelet count >100 x 109/L, hemoglobin > 6,2 mmol/L
  2. Hepatic: Bilirubin within normal range, aspartate transaminase (AST) and alanine transaminase (ALT) <2.5 upper normal lever, albumin > 25 g/L
  3. Renal: creatinine clearance >30 mL/min/1.73m2

     Exclusion Criteria:

     - 1. History of significant gastric or small bowel resection, malabsorption syndrome, or other lack of integrity of the upper gastrointestinal tract that may prevent compliance with oral drug administration 2. Presence of any serious concomitant systemic disorders and/or psychiatric condition incompatible with the study (at the investigator's discretion) 3. Presence of any active infection (at the investigator's discretion). 4. Central nervous system (CNS) disease including epilepsy or altered mental status precluding understanding of the informed consent process and/or completion of the necessary study procedures.

     5. Concurrent use of cationic amphiphilic drugs (see appendix A) including over-the-counter medication.

     6. Use of other investigational drug 7. Allergic reaction to any of the included drugs

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Changes in the profile and concentration of urinary lipids and blood lipids | Blood+urine samples are collected at baseline, at evaluation scans (after 4th and 7th cycles), and at the end of treatment (after 10 Docetaxel cycles, upon progression before 10 cycles, or at study discontinuation). Each cycle is 21 days.
  Measurement of lipid species concentration, focusing on Bis(monoacylglycero)phosphate and lysophospholipids in urine and blood, before, during, and after treatment, compared to PSA levels, radiologic response, and control group results.

SECONDARY OUTCOMES:
radiologic progression-free survival | By comparing with a baseline scan, the treatment effect and disease status will be evaluated with a scan after the 4th and 7th cycles, at end of treatment undtil study completion. Each cycle is 21 days. A patient will receive a maximum of 10 cycles.
  Radiologic progression-free survival is defined as ≥ two new lesions on an 8-week bone scan plus two additional lesions on a confirmatory scan, ≥ two new confirmed lesions on any scan ≥ 9 weeks after enrolment, and/or progression in nodes or viscera on cross-sectional imaging as defined by RECIST 1.1 (see below), or death.
PSA response | PSA response will be monitored during treatment, compared to radiologic response after the 4th and 7th cycles, and at treatment completion (maximum 10 cycles/progression/discontinuation). Each cycle lasts 21 days
  Prostate-Specific Antigen (PSA) Response criteria according to Prostate Cancer Working Group (PCWG3) 3rd edition

CONTACTS AND LOCATIONS:
Overall Officials: Helle Pappot, DMsc, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Department of Oncology 5073, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No